CLINICAL TRIAL: NCT04202588
Title: Gastrointestinal Symptoms Characteristics and Chinese Medicine Patterns in Patients With Functional Gastrointestinal Disorders (FGIDs) in China: a Multicenter Cross-sectional Investigation
Brief Title: A Cross-sectional Investigation on Characteristics of Gastrointestinal Symptoms in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Higher Education Mega Center Branch of Guangdong Provincial Hospital of Chinese Medicine (Unknown); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); Wuhan Hospital of Traditional Chinese Medicine (Other); Hospital of Shanxi University of Traditional Chinese Medicine (Unknown); First Affiliated Hospital of Guizhou University of Traditional Chinese Medicine (Unknown); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Liuzhou Traditional Chinese Medical Hospital (Unknown); Shaanxi Hospital of Traditional Chinese Medicine (Other); Shanghai University of Traditional Chinese Medicine (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Beijing Hospital of Traditional Chinese Medicine Affiliated with Capital Medical University (Unknown); Henan University of Traditional Chinese Medicine (Other); Second Affiliated Hospital of Fujian Traditional Chinese Medical University (Unknown); Inner Mongolia Autonomous Region Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Zhong Lidan, Assistant Professor, Hong Kong Baptist University
Other Study IDs: NationCor-FGID
Record Dates: First submitted 2019-11-25; First posted 2019-12-17 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will conduct a multicenter cross-sectional study to discover symptom characteristics, quality of life, severity of anxiety and depression, status of lactose intolerance and treatment satisfaction of current Chinese Medicine (CM) regimens of outpatients with FGIDs. In the meanwhile, the investigators will also analyze the characters of CM patterns and corresponding elements, then explore the potential relationship between CM patterns and FGIDs' subtypes.

DETAILED DESCRIPTION:
This is a multicenter cross-sectional study to discover symptom characteristics, quality of life, severity of anxiety and depression, status of lactose intolerance and treatment satisfaction of current Chinese Medicine (CM) regimens of outpatients with FGIDs. Afterwards, the investigators will explore the potential relationship between CM patterns and FGIDs' subtypes based on collected information. It is estimated that 4,632 outpatients from 18 centers across China will be recruited. Various demographic and disease-related information will be documented, including name, gender, age, education level, marital status, job category, disease course, medical consultation experience, current CM regimens and rationale, and treatment satisfaction. Patients will also complete a series of scales, containing, Rome IV Diagnostic Questionnaire, Patient-Reported Outcome (PRO) scale, the 36-Item Short Form Survey (SF-36), Hamilton Anxiety Scale (HAMA), Hamilton Depression Scale (HAMD), lactose food frequency questionnaire (Lactose FFQ) and CM pattern scale. The primary outcome will be the symptom characteristics of outpatients with FGIDs. Secondary outcomes include population characteristics of FGID patients (quality of life, emotional status, lactose intolerance status, and satisfaction level of CM interventions), and potential association between CM patterns and FGIDs' subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms onset at least 3 months
* Meet the diagnostic criteria of FGIDs
* Informed consent and ability to read and understand questionnaires

Exclusion Criteria:

* Combined with organic gastrointestinal diseases
* Appearance of gastrointestinal alarm symptoms
* Combined with mental disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients of third-class hospitals across China
Sampling Method: Non-Probability Sample
Enrollment: 4632 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of different subtypes with Functional gastrointestinal disorders (FGIDs) in China | 2 years
  The percentage of the different subtypes with FGIDs by Rome IV Diagnostic Criteria
The health-related quality of life (HRQOL) of outpatients with FGIDs in China | 2 years
  The HRQOL scale contains 36 questions scoring from 0 to 4. Higher score means a worse outcome. The highest total score is 144.

SECONDARY OUTCOMES:
Demographic characteristics of outpatients with FGIDs in China | 2 years
  Including age, gender, education level, marital status and job categories
Quality of life of outpatients with FGIDs in China | 2 years
  36-Item Short Form Survey (SF-36) will be used. Thirty items are contained and each item is scored on a 0 to 100 range. A high score defines a more favorable health state.
HAMA scoring of outpatients with FGIDs in China | 2 years
  Hamilton Anxiety Scale (HAMA) contained and 14 questions scoring form 0 to 4. A high score means a worse anxiety state.
HAMD scoring of outpatients with FGIDs in China | 2 years
  Hamilton Depression Scale (HAMD) contained and 17 questions scoring form 0 to 4. A high score means a worse depression state.
Treatment satisfaction score of CM interventions in outpatients with FGIDs in China | 2 years
  Treatment satisfaction will be evaluated using a single question scoring from 0 to 4. A higher score means worse satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Linda Zhong, Kowloon Tong, Kowloon, Hong Kong